CLINICAL TRIAL: NCT05096611
Title: Efficacy of an Integrated Intervention to Treat Maternal Depression and Children's Behavior Problems: A Transactional Perspective
Brief Title: Attachment and Biobehavioral Catch-up and Depression Treatment
Acronym: ABC+D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A137439; R56MH127032 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-10-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Maternal Depression; Child Behavior Problem

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABC (Active Comparator): Attachment and Biobehavioral Catch-up, 10 weekly sessions that provide parenting support
  Interventions: Behavioral: Attachment and Biobehavioral Catch up
- ABC+D (Experimental): Attachment and Biobehavioral Catch-up plus weekly 5-10 minute videos that additional provide support for mothers' mood, stress, and coping
  Interventions: Behavioral: Attachment and Biobehavioral Catch up Plus Depression Treatment

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch up — ABC is delivered by a trained parent coach. The parent coach provides information about parenting and child development. The focus is on providing support for parents of young children and improving the parent-child relationship.
  Other Names: ABC
  Arms: ABC
Behavioral: Attachment and Biobehavioral Catch up Plus Depression Treatment — ABC+D offers the same 10-sessions of parenting support that is provided by ABC and additionally provides weekly short videos that help mothers develop skills for coping with stress and regulating mood.
  Other Names: ABC+D
  Arms: ABC+D

SUMMARY:
Maternal depression influences the development of children's behavior problems and vice versa; however most interventions singularly address maternal depression or children's behavior problems rather than both. This project assesses the efficacy of an intervention that treats both mothers and children in an integrated manner. Effects are expected to disrupt the reciprocal relations that perpetuate maternal and child mental health problems over time.

DETAILED DESCRIPTION:
The proposed project is a pilot randomized controlled trial to evaluate the effectiveness of an integrated intervention that dually treats maternal depressive symptoms and offspring behavior problems. Families (n = 40 mothers and their 2-to-4 year-old children) will be randomized to receive 10 sessions of ABC or 10 sessions of ABC+D in their home. ABC+D is an expanded version of ABC that additionally treats maternal depressive symptoms using Mothers and Babies adapted for mothers of toddlers. The specific aims of this proposed project are:

Aim 1. Collect preliminary data on the feasibility and acceptability of ABC+D in preparation for a small pilot randomized controlled trial (RCT).

Aim 2. Conduct a small pilot RCT to examine the effectiveness of ABC and ABC+D

Aim 3: Assess the overall acceptability (mother- and provider-rated), appropriateness (mother- and provider-rated), and feasibility (provider-rated) of ABC+D. Mothers will also rate their satisfaction with each session and the degree to which it was helpful, interesting, and comprehensible.

ELIGIBILITY:
Inclusion Criteria:

1. Mothers 18 years of age or older with heightened depressive symptoms as determined by a score of 5 or higher on the Patient Health Questionnaire-9 (PHQ-9)
2. Biological children (of mothers described above) between 2 and 4 years old with heightened behavior problems as determined by a score of at least 3 in at least 1 domain of functioning on the Impairment Rating Scales
3. English- or Spanish-speaking

Exclusion Criteria:

1. Self-reported history of psychosis or active suicidality as defined by self-report of a specific suicide plan or recent attempt
2. Child diagnosis of autism

Min Age: 2 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Score | Baseline to post-intervention. This is an anticipated average of 10 weeks.
  Scores range from 34.5 to 82.3 with higher values indicating more severe symptoms
Change in Early Childhood Screening Assessment score | Baseline to post-intervention. This is an anticipated average of 10 weeks.
  Scores range from 0 to 72 with higher values indicating more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Roubinov, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the NIMH Data Archive (NDA)
Time Frame: Data from this clinical trial require significant processing after the completion of data collection. We will submit a clean dataset after the final data lock.
Access Criteria: Researchers will the appropriate qualifications can request the dataset via the NIMH Data Archive Platform.